CLINICAL TRIAL: NCT05376826
Title: A Study to Assess the Effectiveness of Nurse-led Physical Therapy in Terms of Patient Competency, Patient Engagement and Physical Performance Among CLD Patients With Physical Frailty.
Brief Title: Effectiveness of Nurse-led Physical Therapy in Terms of Patient Competency, Patient Engagement and Physical Performance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ILBS-CLD-02
Record Dates: First submitted 2021-10-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-10

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: Patient Competency; Patient engagement; Physical Performance; CLD; MELD
MeSH Terms: conditions — Fibrosis; Patient Participation

STUDY DESIGN:
Intervention Model Description: Pre-test - Post test Control group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefrail and Frail CLD Patients (Experimental): Nurse- led Physical Therapy include Video based range of Motion Exercises for 10-20 min.
  Interventions: Behavioral: Nurse Led Physical Therapy
- Control Group (No Intervention): Routine Interventions

INTERVENTIONS:
Behavioral: Nurse Led Physical Therapy — Nurse Led Physical Therapy in Form of Range of Motion Exercises
  Arms: Prefrail and Frail CLD Patients

SUMMARY:
Due to Prolonged diseased Condition, Patients are not able to care for themselves and even avoid movement their range of motion is limited which may develop frailty among Liver disease Patients.

This Study aims at assessing Engagement, Competency and Physical Performance of Physical Frail Chronic Liver disease Patients before and after Nurse led Physical therapy.

Besides these Parameters effect of Intervention on Physical frailty will also be assessed.

DETAILED DESCRIPTION:
Research Approach: Quantitative Study Research design: Quasi Experimental Research design ( Pre-test - Post test Control group design) Setting: Study is planned on OPD patients of ILBS, New Delhi. Sampling Technique: Random Allocation in Experiment and Control group after matching for age and gender Sample size: 80 Patients Variables: Independent variable- Nurse-led Physical therapy Dependent Variable- Patient Competency, Patient Engagement, Physical Performance.

ELIGIBILITY:
Inclusion Criteria:

* Prefrail and Frail CLD Patients (MELD <24)
* Follow up of Prefrail and Frail CLD Patients (MELD<24)
* Participants willing for Research

Exclusion Criteria:

* Frail Patients who are bedridden
* presence of hepatopulmonary disease
* Presence of neurological defects
* Previous history of Liver Transplantation
* Severe COPD, Heart Failure

Ages: 20 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Patient Competency by patient Competency Scale at 1 week | 1 week
  Compare Patient Competency using patient Competency Scale. The total score of this scale ranges from 0-84 with minimum score 28 and maximum score 84. Higher scores mean a highly competent score.

SECONDARY OUTCOMES:
Patient Engagement by Patient Engagement Scale at 1 week | 1 week
  Patient Engagement using Patient Engagement Scale. The total score of this scale ranges from 10-40 with minimum score 10 and maximum score 40. Higher scores mean a highly engaged.
Physical Performance by six minute walk test at 1 week | 1 week
  Physical Performance using six minute walk test in Physically Frail Chronic Liver disease patients before and after Physical Therapy. The distance covered measures physical performance, where distance more than 300 meter means normal physical performance and less than or equal to 300 meter means low physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Sonam Ms Kumari, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Sonam Kumari, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No